CLINICAL TRIAL: NCT00534963
Title: Optimal Catheter Placement During Sonohysterography: A Randomized Clinical Trial Comparing Cervical to Uterine Placement
Brief Title: Optimal Catheter Placement During Sonohysterography: Comparison of Cervical to Uterine Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-2004-0066
Record Dates: First submitted 2007-09-23; First posted 2007-09-26 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Catheter Placement and Perceived Pain
Keywords: sonohysterography, catheter placement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: cervical vs. uterine placement of balloon catheter

SUMMARY:
The primary objective of this investigation was to evaluate if the location of placement of the SIS balloon into either the uterine cavity or the cervical canal affected discomfort perceived during the examination.

DETAILED DESCRIPTION:
The use of sonography combined with intrauterine saline instillation, termed sonohysterography

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing SIS for diagnostic uterine cavity evaluation at our university's Reproductive Endocrine Infertility Program.

Exclusion Criteria:

* previous hysterectomy, current pregnancy, active PID, patulous or stenotic cervical os noted on previous history or physical exam.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-12; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Measure: perceived discomfort | during sonohysterography procedure

SECONDARY OUTCOMES:
Measure: Time required to perform procedure; Measure: Volume of media required to perform procedure | during sonohysterography procedure

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindheim, MD, Principal Investigator — University of Wisconsin Department of Reproductive Endocrinology and Infertility

REFERENCES:
- [Derived] Spieldoch RL, Winter TC, Schouweiler C, Ansay S, Evans MD, Lindheim SR. Optimal catheter placement during sonohysterography: a randomized controlled trial comparing cervical to uterine placement. Obstet Gynecol. 2008 Jan;111(1):15-21. doi: 10.1097/01.AOG.0000295865.93719.3f. PMID 18165388